CLINICAL TRIAL: NCT00021710
Title: Motor Learning: Behavioral and Physiologic Studies in Normal Volunteers and Stroke Patients
Brief Title: Motor Learning in Stroke Patients and Healthy Volunteers
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010220; 01-N-0220
Record Dates: First submitted 2001-08-02; First posted 2001-08-03 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-06

CONDITIONS: Stroke; Healthy
Keywords: Stroke; Learning; Plasticity; Motor; Rehabilitation; Premotor; Normal Control; Healthy Volunteer; HV; Motor Learning
MeSH Terms: conditions — Stroke

SUMMARY:
This study will try to elucidate learning processes associated with motor training in the weak arm of stroke patients compared with healthy controls. Results from previous clinical trials indicate that training may enhance motor function in healthy volunteers, and perhaps also in stroke patients, even more than 1 year after the stroke. Normal, healthy volunteers and stroke patients 18 years of age and older may be eligible for this study.

Study subjects will have a physical examination and participate in 6 additional clinic visits-training and testing sessions on study days 1, 2, 3, 4 and 5, and a final testing session on day 12. During these sessions, they will perform a series of motor tasks, including writing, picking up objects, turning cards, stacking checkers and moving cans, which will be timed and videotaped. Each session will be divided into blocks of 10 trials for each task, separated by 2-minute rest periods.

Before and after training on days 1, 2, 5 and 12, subjects will have transcranial magnetic stimulation (TMS) to determine brain changes associated with learning a motor task. For this procedure, the patient is seated in a comfortable chair, and an insulated wire coil is placed on the scalp or skin. A brief electrical current is passed through the coil, creating a magnetic pulse that stimulates the brain. These pulses generate very small electrical currents in the brain cortex, briefly disrupting the function of the brain cells in the stimulated area. The stimulation may cause muscle twitching or tingling in the scalp, face, or limb. During the stimulation, the subject may be asked to slightly tense certain muscles or perform other simple actions.

Electrical nerve stimulation and electromyography will be done to record muscle responses to stimulation. A nerve is stimulated by placing wires on the skin over the nerve and passing a brief electrical current between the wires. Electromyography involves taping metal electrodes to the skin over the muscle.

Before and after each session, subjects' muscle strength will be tested with a pinch gauge. They will also be asked to make a mark on a line drawn on paper, to rate their test performance and levels of attentiveness and fatigue.

DETAILED DESCRIPTION:
The purpose of this protocol is to characterize dynamics of motor learning over a 5-day period in chronic stroke patients relative to healthy age-matched controls. Motor learning will be assessed by improvements in the Jebsen-Taylor test, a validated tool widely used in rehabilitation that measures upper extremity function. Additionally, we intend to evaluate changes in the excitability of the primary motor cortex associated with learning using transcranial magnetic stimulation.

ELIGIBILITY:
INCLUSION CRITERIA FOR HEALTHY VOLUNTEERS

Age: 18 years to 100 years

Normal physical and neurological examinations

EXCLUSION CRITERIA FOR HEALTHY VOLUNTEERS

Contraindications for transcranial magnetic stimulation: pacemaker, implanted medical pump, metal plate in skull, metal objects inside the eye or skull, history of seizures

INCLUSION CRITERIA FOR STROKE PATIENTS

Age: 18 years to 100 years

Single ischemic or hemorrhagic hemispheric stroke at least one year before enrollment in study, confirmed by neuroimaging studies (computerized tomography or magnetic resonance imaging).

Ability to perform the Jebsen-Taylor test.

EXCLUSION CRITERIA FOR STROKE PATIENTS

More than one stroke.

Other brain lesions (i.e., traumatic brain injury, brain tumor) or neurological problems (i.e., multiple sclerosis, dementia, Parkinson's disease)

Depression or poor motivational capacity

Serious cognitive deficits (defined as equivalent to a mini-mental state exam score of 20 or less).

Inability to understand instructions for the Jebsen-Taylor test.

Uncontrolled medical problems including cardiovascular disease, severe rheumatoid arthritis, active joint deformity of arthritic origin, active cancer or renal disease, any kind of end-stage pulmonary or cardiovascular disease, uncontrolled epilepsy

Contraindications for transcranial magnetic stimulation: pacemaker, implanted medical pump, metal plate in skull, metal objects inside the eye or skull, history of seizures

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 78
Dates: Start 2001-07; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Boyd LA, Winstein CJ. Implicit motor-sequence learning in humans following unilateral stroke: the impact of practice and explicit knowledge. Neurosci Lett. 2001 Jan 26;298(1):65-9. doi: 10.1016/s0304-3940(00)01734-1. PMID 11154837
- [Background] Bridgers SL, Delaney RC. Transcranial magnetic stimulation: an assessment of cognitive and other cerebral effects. Neurology. 1989 Mar;39(3):417-9. doi: 10.1212/wnl.39.3.417. PMID 2927652
- [Background] Butefisch C, Hummelsheim H, Denzler P, Mauritz KH. Repetitive training of isolated movements improves the outcome of motor rehabilitation of the centrally paretic hand. J Neurol Sci. 1995 May;130(1):59-68. doi: 10.1016/0022-510x(95)00003-k. PMID 7650532